CLINICAL TRIAL: NCT01330160
Title: Characterization of Clinical, Biological, Morphological and Pharmacological Factors Influencing Occurrence of Dementia or Cognitive Disorders After Stroke
Brief Title: Study of Factors Influencing Post-stroke Dementia
Acronym: strokdem
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2008_42/0907; 2008/API1901 (Other Grant/Funding Number: PHRC); 2009-A00141-56 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2010-10-01; First posted 2011-04-06 (Estimated); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Cerebrovascular Disorders; Dementia
Keywords: stroke; Brain ischemia; Intracranial hemorrhage; Dementia, Vascular; Alzheimer's disease
MeSH Terms: conditions — Cerebrovascular Disorders; Dementia; Stroke; Brain Ischemia; Intracranial Hemorrhages; Dementia, Vascular; Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — standard biological parameters (ionogram, blood count, glycemia, lipids, renal function, vitamin B12, thyroid hormones, homocysteinemia), specialized biology (inflammation, oxidative, vascular biomarkers ; amyloid and tau markers), genotype (apolipoprotein E, apolipoprotein C, kinesin, Angiotensin Converting Enzyme...).
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- cohort of stroke patients: patients, over 40 years old and without dementia, displaying an hemorrhagic or an ischemic stroke, with a sus-tentorial localization, and included 72h before the onset of symptoms

SUMMARY:
If the risk of dementia occurrence after stroke is well known, few data exist about the factors influencing positively or negatively the developement of cognitive disorders or dementia. The aim of the study is so to determine prospectively the clinical, biological, lesional and pharmacological factors associated with post-stroke dementia by the long-term follow-up of a stroke patient cohort.

DETAILED DESCRIPTION:
The STROKDEM study is based on the 5-year prospective follow-up of a population of 1100 stroke patients without dementia. At inclusion in the cohort, main antecedents and risk factors, previous treatment and lifestyle, initial severity and etiology are recorded. Biological samples (for standard ans specialized analyses) and MRI are performed at 72h after stroke occurrence. Thereafter, patients are regularly (6 months, 12 months, 36 months, 60 months) examined for clinical and cognitive assessment with biological samples and Magnetic Resonance Imaging. Patients with dementia will be compared to patients without stroke to identify, by logistic regression analysis and Cox model, the factors associated with dementia occurrence.

ELIGIBILITY:
Inclusion Criteria:

* patients > 40 years olds
* hemispheric stroke
* stroke dating from less 72h
* IQ-code < 64
* patient (or his family) given an informed consent

Exclusion Criteria:

* non hemispheric stroke
* malformative intracranial hemorrhage
* traumatic intracranial hemorrhage
* subarachnoidal hemorrhage
* contra-indication to MRI
* patients unable to answer to cognitive battery

Ages: 40 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients without dementia displaying an hemispheric ischemic or hemorrhagic stroke hospitalized during the 72h following the beginning of stroke
Sampling Method: Non-Probability Sample
Enrollment: 229 (Actual)
Dates: Start 2010-02-27 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
dementia occurrence | 60 months
  This evaluation will be based on a neurological and general clinical examination, and on the evaluation of activities of daily life using the Instrumental Activities Daily Life scale after an interview with the patient and his/her family.

SECONDARY OUTCOMES:
dementia occurrence and cognitive impairment | 6 months
  This evaluation will be based on a neurological and general clinical examination, and on the evaluation of activities of daily life using the Instrumental Activities Daily Life scale after an interview with the patient and his/her family.
  Impairment of some tests of cognitive battery without significant impairment in activities of daily living
dementia occurrence and cognitive impairment | 12 months
  This evaluation will be based on a neurological and general clinical examination, and on the evaluation of activities of daily life using the Instrumental Activities Daily Life scale after an interview with the patient ans his/her family.
  Impairment of some tests of cognitive battery without significant impairment in activities of daily living
dementia occurence and cognitive impairment | 36 months
  This evaluation will be based on a neurological and general clinical examination, and on the evaluation of activities of daily life using the Instrumental Activities Daily Life scale after an interview with the patient ans his/her family.
  Impairment of some tests of cognitive battery without significant impairment in activities of daily living
cognitive impairment | 36 months
  Impairment of some tests of cognitive battery without significant impairment in activities of daily living

CONTACTS AND LOCATIONS:
Overall Officials: Regis Bordet, MD PhD, Study Chair — Lille University Hospital
Locations (4):
- France (4):
  - Amiens University Hospital, Amiens
  - Caen University Hospital, Caen
  - Lille University Hospital, Lille
  - Rouen University Hospital, Rouen

REFERENCES:
- [Result] Deplanque D, Bastide M, Bordet R. Transient Ischemic Attack and Minor Stroke: Definitively Not So Harmless for the Brain and Cognitive Functions. Stroke. 2018 Feb;49(2):277-278. doi: 10.1161/STROKEAHA.117.020013. Epub 2018 Jan 4. No abstract available. PMID 29301969
- [Derived] Mazella E, Mendyk AM, Accart B, Borsotto M, Heurteaux C, Bordet R, Mazella J, Dondaine T. Serum sortilin-derived propeptide concentrations as markers of depression in chronic stroke. J Neurol Sci. 2025 May 15;472:123459. doi: 10.1016/j.jns.2025.123459. Epub 2025 Mar 8. PMID 40107034
- [Derived] Ponchel A, Labreuche J, Bombois S, Delmaire C, Bordet R, Henon H. Influence of Medication on Fatigue Six Months after Stroke. Stroke Res Treat. 2016;2016:2410921. doi: 10.1155/2016/2410921. Epub 2016 Jun 19. PMID 27413577